CLINICAL TRIAL: NCT07008079
Title: Flapless Mini-incision Implant Surgery vs Conventional Flap or Flapless Implant Surgery: A Prospective, Randomized, Single Blind, Clinical and Radiographic Study
Brief Title: Flapless Mini-incision Implant Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alaa Emara (Other)
Collaborators: King Saud University (Other)
Responsible Party: Sponsor-Investigator, Alaa Emara, A.Professor, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Flapless mini-incision implant
Record Dates: First submitted 2025-05-19; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: IMPLANTATION; Dental Implant; Dental Implant Placement; Peri-Implant Tissues
Keywords: flapless surgery; mini-incision surgery; peri-implant soft tissue; dental implant

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional flap (Active Comparator): The Standard commonly used surgical flap is used to place the dental implant
  Interventions: Procedure: Conventional flap
- Flapless punch (Experimental): A flapless punch is used to place the dental implants
  Interventions: Procedure: Flapless punch
- Flapless mini-incision (Experimental): A flapless mini incision is used to place the dental implants
  Interventions: Procedure: Flapless mini-incision

INTERVENTIONS:
Procedure: Flapless punch — use of flapless puch surgery to place dental implants
  Arms: Flapless punch
Procedure: Flapless mini-incision — Use of a flapless mini-incision to place a dental implant
  Arms: Flapless mini-incision
Procedure: Conventional flap — Use of a conventional surgical flap to place a dental implant
  Arms: Conventional flap

SUMMARY:
evaluate the clinical efficacy of the flapless mini-incision method compared to conventional flap and flapless punch methods

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with adequate bone height and width at the site of implant 120 placement, and good quality bone to support a primary stability of at least 30 Ncm and D2 bone quality according to Lekholm and Zarb classification), based on preoperative radiographic assessment
* Clinical evidence of optimal periodontal health with no active periodontal disease in adjacent teeth
* No history of systemic illnesses that could affect bone health and wound heal- ing (e.g. uncontrolled diabetes mellitus, osteoporosis, renal osteodystrophy…etc.)
* No history of or requirement for bone grafting and augmentation at the implant site
* Willingness to participate in the study and attend prescribed follow-up appointments

Exclusion Criteria:

* Patients with history of radiation therapy for head and neck cancer
* Patients with history of allergy and hypersensitivity to local anesthetic agents, and biomaterials used in dental implants
* Pregnant women and lactating mothers
* History of smoking (>2 cigarettes per day)
* Patients under treatment with anti-resorptive or anti-neoplastic medication such as bisphosphonates, chemotherapeutic agents, and monoclonal antibodies (e.g. Denosumab

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Pain score | 18 months postoperatively
  Assessment of patient's pain level using Visual Analog Scale (VAS) which would be compared between groups.
  VAS is a visual scale 0 to 10 with 10 the highest pain score and 0 the lowest, the patient is asked to identify the pain level at the different timestops for comparison between groups

SECONDARY OUTCOMES:
Soft-tissue healing | 18 months postoperatively
  Assess the healing of overlaying soft tissue. Check for signs of infection , swelling, dehiscnce or inflammation
Radiographic bone level | 18 months postoperatively
  Assessment of bone level postoperatively. A CBCT is ordered to assess bone density in hounsfeld unitsto assess level of bone maturation. This would then be compared across groups and between different time points to show bone deposition and healing.

CONTACTS AND LOCATIONS:
Locations (1):
- King Saud University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided
We might be sharing our data when needed according to the case